CLINICAL TRIAL: NCT00005398
Title: University of North Carolina Alumni Heart Study
Status: Active, not recruiting | Type: Observational
Sponsor: Duke University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: Pro00013233; R01HL055356 (NIH); P01HL036587 (NIH); R01MH066079 (NIH); 4311
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Coronary Disease; Depression
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Coronary Disease; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1; no experimental groups in this study: Observational cohort study
  Interventions: Other: There is no intervention

INTERVENTIONS:
Other: There is no intervention — No applicable

SUMMARY:
To continue surveillance of the participants in the University of North Carolina Alumni Heart Study, which tests the hypothesis that hostility and related psychosocial factors are involved in the pathogenesis of coronary heart disease.

DETAILED DESCRIPTION:
BACKGROUND:

Prevention of coronary heart disease (CHD) will be enhanced by controlling hypertension, reducing blood cholesterol, maintaining normal weight, increasing physical activity, reducing smoking, and having a healthy diet. Understanding how to achieve these important public health aims requires an understanding of the behavioral factors involved in prevention. Behavioral risk factors remain the single most preventable cause of human illness and suffering. The University of North Carolina Alumni Heart Study is ideally suited to explore the associations between and among these important behavioral risk factors, and to understand how personality, in particular individual differences in hostility and depression act to determine individuals' risk factor behaviors, and to answer important questions about the role of hostility and psychosocial factors in CHD risk during the middle years.

The University of North Carolina Alumni Heart Study (UNCAHS) is a prospective study of the role of psychosocial factors, in particular hostility, in the development of coronary heart disease. The target population is composed of persons who completed the Minnesota Multiphasic Personality Inventory while attending the University of North Carolina in the mid-1960s.

DESIGN NARRATIVE:

Surveillance of the members of the UNC Alumni Heart Study continues for an additional five-year period . Studies continue on how hostility and other psychosocial factors are related to each other and how they contribute to coronary heart disease risk. Data are analyzed in order to test hypotheses about the role of psychosocial factors in weight parameters, dietary practices and the contribution of spouse hostility to coronary risk.

To better understand the dynamic interrelationships of psychosocial and behavioral risk factors of the adult life span, the trajectories of hostility, depression, smoking, body mass, exercise patterns, and alcohol consumption will be mapped using multiple assessments from age 19 to age 60. It is predicted that a significant proportion of the change in risk behavior will be due to trajectories of hostility and depression, operating singly and in combination over time. Tests will be made of the prospective associations of hostility, depression, and other psychosocial variables (e.g., social support and job strain) with coronary events and mortality observed while the cohort is middle-aged. The scope of the psychosocial variables will be broadened to examine individual differences in personality over the life course and dietary practices at midlife in addition to the indicators noted above. The effect of gender on the natural history of coronary disease and coronary risk profiles in women will be examined by monitoring changes in menopausal status, and patterns of hormone replacement therapy use among women during midlife and the associations of these factors with the other risk indicators.

ELIGIBILITY:
No eligibility criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: participants in the University of North Carolina Alumni Heart Study
Sampling Method: Non-Probability Sample
Enrollment: 6340 (Actual)
Dates: Start 1996-05; Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Coronary Heart Disease | approximately 30 years
  This is a descriptive cohort study

CONTACTS AND LOCATIONS:
Overall Officials: Ilene C. Siegler, PhD, MPH, Principal Investigator — Duke University
Locations (1):
- Duke University, Behavioral Medicine Research Center, Durham, North Carolina, United States

REFERENCES:
- [Background] Brummett BH, Barefoot JC, Feaganes JR, Yen S, Bosworth HB, Williams RB, Siegler IC. Hostility in marital dyads: associations with depressive symptoms. J Behav Med. 2000 Feb;23(1):95-105. doi: 10.1023/a:1005424405056. PMID 10749013
- [Background] Barefoot JC, Heitmann BL, Helms MJ, Williams RB, Surwit RS, Siegler IC. Symptoms of depression and changes in body weight from adolescence to mid-life. Int J Obes Relat Metab Disord. 1998 Jul;22(7):688-94. doi: 10.1038/sj.ijo.0800647. PMID 9705031
- [Background] Bastian LA, Couchman GM, Rimer BK, McBride CM, Feaganes JR, Siegler IC. Perceptions of menopausal stage and patterns of hormone replacement therapy use. J Womens Health. 1997 Aug;6(4):467-75. doi: 10.1089/jwh.1997.6.467. PMID 9279835
- [Background] Luecken LJ, Suarez EC, Kuhn CM, Barefoot JC, Blumenthal JA, Siegler IC, Williams RB. Stress in employed women: impact of marital status and children at home on neurohormone output and home strain. Psychosom Med. 1997 Jul-Aug;59(4):352-9. doi: 10.1097/00006842-199707000-00003. PMID 9251153
- [Background] Herbst JH, McCrae RR, Costa PT Jr, Feaganes JR, Siegler IC. Self-perceptions of stability and change in personality at midlife: the UNC Alumni Heart Study. Assessment. 2000 Dec;7(4):379-88. doi: 10.1177/107319110000700406. PMID 11151963
- [Background] Costa PT Jr, Herbst JH, McCrae RR, Siegler IC. Personality at midlife: stability, intrinsic maturation, and response to life events. Assessment. 2000 Dec;7(4):365-78. doi: 10.1177/107319110000700405. PMID 11151962
- [Background] Siegler IC, Brummett BH. Associations among NEO personality assessments and well-being at midlife: facet-level analyses. Psychol Aging. 2000 Dec;15(4):710-4. doi: 10.1037//0882-7974.15.4.710. PMID 11144330
- [Background] Brummett BH, Maynard KE, Haney TL, Siegler IC, Barefoot JC. Reliability of interview-assessed hostility ratings across mode of assessment and time. J Pers Assess. 2000 Oct;75(2):225-36. doi: 10.1207/S15327752JPA7502_4. PMID 11020141
- [Background] McPherson RS, Feaganes JR, Siegler IC. Measurement of dietary intake in the UNC Alumni Heart Study. University of North Carolina. Prev Med. 2000 Jul;31(1):56-67. doi: 10.1006/pmed.2000.0679. PMID 10896844
- [Background] Barefoot JC, Gronbaek M, Feaganes JR, McPherson RS, Williams RB, Siegler IC. Alcoholic beverage preference, diet, and health habits in the UNC Alumni Heart Study. Am J Clin Nutr. 2002 Aug;76(2):466-72. doi: 10.1093/ajcn/76.2.466. PMID 12145024
- [Background] Siegler IC, Bastian LA, Steffens DC, Bosworth HB, Costa PT. Behavioral medicine and aging. J Consult Clin Psychol. 2002 Jun;70(3):843-51. doi: 10.1037//0022-006x.70.3.843. PMID 12090387
- [Background] Bosworth HB, Siegler IC. Terminal change in cognitive function: an updated review of longitudinal studies. Exp Aging Res. 2002 Jul-Sep;28(3):299-315. doi: 10.1080/03610730290080344. PMID 12079580
- [Background] Vitaliano PP, Scanlan JM, Zhang J, Savage MV, Hirsch IB, Siegler IC. A path model of chronic stress, the metabolic syndrome, and coronary heart disease. Psychosom Med. 2002 May-Jun;64(3):418-35. doi: 10.1097/00006842-200205000-00006. PMID 12021416
- [Background] Surwit RS, Williams RB, Siegler IC, Lane JD, Helms M, Applegate KL, Zucker N, Feinglos MN, McCaskill CM, Barefoot JC. Hostility, race, and glucose metabolism in nondiabetic individuals. Diabetes Care. 2002 May;25(5):835-9. doi: 10.2337/diacare.25.5.835. PMID 11978677
- [Background] Brummett BH, Barefoot JC, Vitaliano PP, Siegler IC. Associations among social support, income, and symptoms of depression in an educated sample: the UNC Alumni Heart Study. Int J Behav Med. 2003;10(3):239-50. doi: 10.1207/s15327558ijbm1003_04. PMID 14525719
- [Background] Siegler IC, Costa PT, Brummett BH, Helms MJ, Barefoot JC, Williams RB, Dahlstrom WG, Kaplan BH, Vitaliano PP, Nichaman MZ, Day RS, Rimer BK. Patterns of change in hostility from college to midlife in the UNC Alumni Heart Study predict high-risk status. Psychosom Med. 2003 Sep-Oct;65(5):738-45. doi: 10.1097/01.psy.0000088583.25140.9c. PMID 14508014
- [Background] Brummett BH, Siegler IC, McQuoid DR, Svenson IK, Marchuk DA, Steffens DC. Associations among the NEO Personality Inventory, Revised and the serotonin transporter gene-linked polymorphic region in elders: effects of depression and gender. Psychiatr Genet. 2003 Mar;13(1):13-8. doi: 10.1097/00041444-200303000-00002. PMID 12605095
- [Background] Boyle SH, Williams RB, Mark DB, Brummett BH, Siegler IC, Barefoot JC. Hostility, age, and mortality in a sample of cardiac patients. Am J Cardiol. 2005 Jul 1;96(1):64-6. doi: 10.1016/j.amjcard.2005.02.046. PMID 15979435
- [Background] Applegate KL, Keefe FJ, Siegler IC, Bradley LA, McKee DC, Cooper KS, Riordan P. Does personality at college entry predict number of reported pain conditions at mid-life? A longitudinal study. J Pain. 2005 Feb;6(2):92-7. doi: 10.1016/j.jpain.2004.11.001. PMID 15694875
- [Background] Brummett BH, Boyle SH, Siegler IC, Williams RB, Mark DB, Barefoot JC. Ratings of positive and depressive emotion as predictors of mortality in coronary patients. Int J Cardiol. 2005 Apr 20;100(2):213-6. doi: 10.1016/j.ijcard.2004.06.016. PMID 15823627
- [Background] Brummett BH, Mark DB, Siegler IC, Williams RB, Babyak MA, Clapp-Channing NE, Barefoot JC. Perceived social support as a predictor of mortality in coronary patients: effects of smoking, sedentary behavior, and depressive symptoms. Psychosom Med. 2005 Jan-Feb;67(1):40-5. doi: 10.1097/01.psy.0000149257.74854.b7. PMID 15673622